CLINICAL TRIAL: NCT02525705
Title: Frequency of Occurrence of Dumping Syndrome After Operation of Esophageal Atresia Type III
Brief Title: Dumping Syndrome After Operation of Esophageal Atresia Type III
Acronym: DUMPING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009_42/1004; 2010-A00217-32 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Oesophageal Atresia; Dumping Syndrome
Keywords: infants; oesophageal atresia; dumping syndrome; prevalence; Type III and IV; Oral glucose tolerance test; early hyperglycemia; late hypoglycemia
MeSH Terms: conditions — Esophageal Atresia; Dumping Syndrome; Hyperglycemia | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Every EA patients (Experimental): This is a one group interventional study. Every patient is included in the same arm.
  Interventions: Biological: Oral Glucose

INTERVENTIONS:
Biological: Oral Glucose — 1.75g/kg of glucose is orally taken by the patient. Capillary glycemia is systematically realised before ingestion (H0) and after 30, 60, 90, 120, 180 and 240 min and/or if clinical signs of hypoglycemia are presented by the patient.

SUMMARY:
The purpose of this study is to evaluate the prevalence at 3.5 months of age of dumping syndrome in children operated at birth for oesophageal atresia type III et IV.

DETAILED DESCRIPTION:
Consecutive patients with type III and IV oesophageal atresia that are born in 8 different centers in France and Sydney (Australia) are included in the study, if willing. As soon as they weigh more than 4.150kg and if they are still younger than 3.5 months, an Oral Glucose Tolerance Test (OGTT) is performed. Glycemia and insulinemia are monitored every 30 minutes from intake to 240 minutes. Clinical signs that are presented are noted. If early hyperglycemia or late hypoglycemia are biologically or clinically observed, ascarbose treatment is initiated.

ELIGIBILITY:
Inclusion Criteria:

* New born less than 3.5 months or age corrected for premature new born
* Weight ≥ 4, 150 kg
* Esophageal atresia (EA) type III or IV
* EA Surgery between May 2013 and June 2016
* Stop of prokinetic treatment > 72 h before OGTT
* Information and consent of parents
* Patients with health insurance

Exclusion Criteria:

* Age > 3.5 months
* Weight < 4.150 kg
* Other types of EA
* Dumping syndrom from other origin: microgastria, dysautonomia, small intestine surgery
* Other pathology that can modify glycemia: neonatal diabete, hyperinsulinism
* Treatment that can modify gastric motility: domperidone, erythromycin, baclofen that hasn't been stopped in the 72h before OGTT
* Absence of consent
* Patient judiciary protected
* Simultaneous participation to another clinical trial
* No health insurance

Max Age: 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2011-06-14 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Early hyperglycemia during Oral Glucose Tolerance Test (OGTT) | up to 240 min
  Hypoglycemia : glycemia < 0,6 g/L
Late hypoglycemia during OGTT | up to 240 min
  Hyperglycemia : > 1,8g/L from H0 to 30 min after oral intake, > 1.7 between 1 and 2 h ours, > 1.4 between 2 and 3 h
  , > 1, 26 after 3 h

SECONDARY OUTCOMES:
Clinical signs presenting consequently to OGTT | continuous monitoring during 240 minutes
  frequent clinical reflux (>3/day), suspicion of esophagitis (pain while eating), colics, post-prandial diarrhea (liquid stools in the first hour after meal), abdominal pain, flatulence, pallor, hypotonia, agitation, convulsions, somnolence, sweat
Associated pathologies | 1 day
  neurologic, extremities, ribbs and vertebrales, genito-urinary, renal, cardiovascular, ano-rectal, microgastria and others. Syndromic associations are also noted, as VACTERL and charge syndroms.
Surgery details | 1 day
  postponed anastomosis, difficulty or tension in the suture, colic or gastric plasty if needed, tracheoscopy realisation, visualisation or damage of the X nerve, observation of a microgastria during surgery, other relevant informations of surgery
Post-surgery complications | 1 day
  anastomotic leakage, mediastinitis

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Michaud, MD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - Hôpital Pellegrin - Hôpital d'Enfants,, Bordeaux
  - CHU Grenoble, Grenoble
  - Hôpital Jeanne de Flandre CHRU, Lille
  - Hôpital Edouard Herriot,Unité d'Hépatogastroentérologie et Nutrition Pédiatriques, Lyon
  - CHU Nantes, Nantes
  - AP-HP, Hôpital Necker, Paris
  - Hôpital Robert Debré ,Service de chirurgie viscérale et urologique, Paris
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Hôpital Enfant, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bufler P, Ehringhaus C, Koletzko S. Dumping syndrome: a common problem following Nissen fundoplication in young children. Pediatr Surg Int. 2001 Jul;17(5-6):351-5. doi: 10.1007/s003830000525. PMID 11527163
- [Result] Samuk I, Afriat R, Horne T, Bistritzer T, Barr J, Vinograd I. Dumping syndrome following Nissen fundoplication, diagnosis, and treatment. J Pediatr Gastroenterol Nutr. 1996 Oct;23(3):235-40. doi: 10.1097/00005176-199610000-00006. PMID 8890072
- [Result] Zung A, Zadik Z. Acarbose treatment of infant dumping syndrome: extensive study of glucose dynamics and long-term follow-up. J Pediatr Endocrinol Metab. 2003 Jul-Aug;16(6):907-15. doi: 10.1515/jpem.2003.16.6.907. PMID 12948306
- [Result] Ng DD, Ferry RJ Jr, Kelly A, Weinzimer SA, Stanley CA, Katz LE. Acarbose treatment of postprandial hypoglycemia in children after Nissen fundoplication. J Pediatr. 2001 Dec;139(6):877-9. doi: 10.1067/mpd.2001.119169. PMID 11743518
- [Result] Michaud L, Sfeir R, Couttenier F, Turck D, Gottrand F. Dumping syndrome after esophageal atresia repair without antireflux surgery. J Pediatr Surg. 2010 Apr;45(4):E13-5. doi: 10.1016/j.jpedsurg.2010.01.016. PMID 20385264
- [Result] Holschneider P, Dubbers M, Engelskirchen R, Trompelt J, Holschneider AM. Results of the operative treatment of gastroesophageal reflux in childhood with particular focus on patients with esophageal atresia. Eur J Pediatr Surg. 2007 Jun;17(3):163-75. doi: 10.1055/s-2007-965087. PMID 17638154
- [Derived] Aumar M, Gottrand F, Chalouhi C, Blanc S, Thomassin N, Piloquet H, Gastineau S, Schneider A, Krishnan U, Duvoisin G, Turck D, Coopman S, Michaud L. Frequency of Abnormal Glucose Tolerance Test Suggestive of Dumping Syndrome Following Oesophageal Atresia Repair. J Pediatr Gastroenterol Nutr. 2020 Jun;70(6):820-824. doi: 10.1097/MPG.0000000000002651. PMID 32443041